CLINICAL TRIAL: NCT06329661
Title: A Multi-center, Randomized, Double-masked, Controlled Clinical Trial to Evaluate the Corneal Endothelial Health of Dry Eye Disease Subjects Treated With Cyclosporine Ophthalmic Solution, 0.1%
Brief Title: A Clinical Trial to Evaluate the Corneal Endothelial Health of DED Subjects Treated With Cyclosporine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYS-007
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclosporine ophthalmic solution, 0.1% (VEVYE) (Active Comparator): Cyclosporine ophthalmic solution, 0.1%; 12 months
  Interventions: Drug: Cyclosporine ophthalmic solution, 0.1%
- Saline solution, 0.6% (Placebo Comparator): Saline solution, 0.6%; 12 months
  Interventions: Drug: Saline solution, 0.6%

INTERVENTIONS:
Drug: Cyclosporine ophthalmic solution, 0.1% — Colorless and clear opthalmic solution containing 0.1% Cyclosporine
  Other Names: VEVYE
  Arms: Cyclosporine ophthalmic solution, 0.1% (VEVYE)
Drug: Saline solution, 0.6% — Colorless and clear sodium chloride solution (0.6%)
  Arms: Saline solution, 0.6%

SUMMARY:
The objective of this trial is to evaluate the effect of cyclosporine ophthalmic solution, 0.1% on corneal endothelial cell health in comparison to a hypotonic saline solution in subjects with Dry Eye Disease (DED)

DETAILED DESCRIPTION:
The effect of cyclosporine ophthalmic solution, 0.1% on corneal endothelial cell density (cells/mm²) will be evaluated in comparison to a hypotonic saline solution in subjects with DED after 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a subject reported history of dry eye disease (DED) in both eyes
* Be able and willing to follow instructions, including participation in all trial assessments and visits.

Exclusion Criteria:

* Be a woman who is pregnant, nursing, or planning a pregnancy;
* Unwillingness to submit a urine pregnancy test at screening and the last visit (or early termination visit) if of childbearing potential, or unwillingness to use acceptable means of birth control
* Clinically significant slit-lamp findings or abnormal lid anatomy at screening
* Ocular/periocular malignancy
* History of herpetic keratitis
* Have any primary or secondary corneal endothelial disorder such as Fuchs dystrophy or other endothelial dystrophy, significant guttata
* Ongoing ocular or systemic infection at screening or baseline
* Presence of uncontrolled systemic diseases
* Presence of known allergy and/or sensitivity to the study drug or its components
* Intraocular surgery or ocular laser surgery or significant trauma within 365 days before Visit 1, or have any planned ocular surgeries during the trial period;
* Have a known allergy or sensitivity to the IMP or its components
* Have a condition or be in a situation which the Investigator feels may put the subject at significant risk, may confound the trial results, or may interfere with the subject's participation in the trial significantly.
* Randomized in a previous CyclASol trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in corneal ECD | 12 months
  ECD measured as count/mm2 using specular microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Krösser, PhD, Study Director — Novaliq GmbH
Locations (6):
- United States (6):
  - CYS-007 Investigational Site, Newport Beach, California
  - CYS-007 Investigational Site, Torrance, California
  - CYS-007 Investigational Site, Garner, North Carolina
  - CYS-007 Investigational Site, Shelby, North Carolina
  - CYS-007 Investigational Site, Cranberry Township, Pennsylvania
  - CYS-007 Investigational Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No